CLINICAL TRIAL: NCT06584500
Title: Analysis of the Effect of Dry Needling on the Pelvitrochanteric Musculature on the Potential Contraction of the Gluteus Medius in Patients with Greater Trochanteric Pain Syndrome: Protocol for a Randomized Clinical Trial. Pilot Study
Brief Title: Effect of Dry Needling on Gluteus Medius Contraction in Greater Trochanteric Pain Syndrome: a Pilot RCT Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Teresa Suárez del Villar Estéfano, María Teresa Suárez del Villar Estéfano, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEIM/2024/4/103
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Greater Trocantheric Pain Syndrome
Keywords: greater trochanteric pain syndrome, potential contraction, dry needling, gluteus medius.
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E Group (Experimental): Experimental group which receives real dry needling
  Interventions: Other: Dry needling
- C Group (Sham Comparator): Control group which receives sham dry needling
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Other: Dry needling — Dry needling will be performed on the pelvitrochanteric musculature, targeting those muscles where the patient reports mechanical hyperalgesia points upon palpation that reproduce familiar and recognizable pain. No more than 3 different muscles will be treated, and no more than 2 needles will be used per muscle to reduce irritability. The Gluteus Medius muscle will be needled in all patients, and the Gluteus Minimus, Tensor Fasciae Latae (TFL), Piriformis, and obturator muscles will also be examined.
  Dry needling will be performed using monofilament needles of different sizes, 0.30mm x 7.5mm, 6mm, and 4mm (AGUPUNT, APS®), depending on the muscle being treated."
  During the dry needling procedure, an attempt will be made to provoke a local twitch response (LTR). Once achieved, the needle will be manipulated with rapid in-and-out movements in different directions until 4 to 6 LTRs are obtained, or if the participant verbally requests the intervention to stop.
  Arms: E Group
Other: Sham Dry Needling — The intervention protocol for sham dry needlig will be just as to the real dry needling procedure, but instead of inserting the needle into the muscle, the needle is manipulated to touch the skin without penetrating it. This may involve the use of retractable needles or simply making contact with the skin
  Arms: C Group

SUMMARY:
Grater trochanteric pain syndrome is a hip related pathology that causes lateral hip pain and lack of strength in abductor muscles such as the gluteus medius, which hinders functional activities and daily life, such as standing, walking, sleeping on the affected side... Lack of strength and eccentric control of the gluteus medius may be related to the apparition of myofascial trigger points that are susceptible to treatment with dry needling.

In this study, two groups of patients with greater trochanteric pain syndrome will be treated with dry needling, some of them with real dry needling, and others with sham dry needling. Ultrasound will be used to assess whether real dry needling in the pelvitrochanteric musculature improves the potential contraction of the gluteus medius, in relation to a baseline measurement and to sham dry needling.

This study is a randomised clinical trial protocol, pilot study, so there will be no previous references for the sample of both study groups. 3 dry needling interventions will be performed in 3 consecutive weeks, leaving 1 week between each intervention. Data will be collected for the variables to be investigated (potential contraction, pain, function, strength…) before the first intervention, after each intervention, 1 month after the last intervention and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Lateral hip pain lasting more than 3 months.
* Greater trochanteric pain syndrome compatible with changes on MRI.
* Clinical examination correlation: one of the following tests must be positive: FADER test, FABER test, hip adduction (ADD) test in side-lying position (DL), isometric contraction test in the ADD position, or single-leg stance test for 30 seconds.
* Pain/sensitization upon palpation of the trochanter.

Exclusion Criteria:

* Radicular pain due to lumbar pathology.
* Osteoarthritis.
* Pelvic pathology that could refer pain to the hip.
* Needle phobia.
* Hip injection performed less than 6 months ago.
* Dry needling performed less than 1 month ago.
* Surgery or pathology of the lower limb that prevents single-leg support.
* Systemic diseases that could interfere with the pathological process.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-09-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Potential Contraction with M-Mode | From enrollment to the end of treatment at 4 months
  The primary variable in this study will measure the potential contraction of the gluteus medius. This variable will be assessed using a Sonoscape E2 ultrasound machine with a 5 cm linear probe and the highest scanning speed. The probe will be positioned at the midpoint of the line connecting the anterior and posterior superior iliac spines. In longitudinal scanning, M-mode will be placed cranially to the hip joint capsule. Thickness will be measured from the inner surface of the fascial borders, with the unit of measurement in millimeters (mm). The contraction potential will be the difference between the thickness of the gluteus medius at rest and the thickness at 80% of the maximum voluntary isometric contraction.

SECONDARY OUTCOMES:
WOMAC hip scale | From enrollment to the end of treatment at 4 months
  This is a scale validated in Spanish to measure disability. Barratt et al. recommend the use of condition-specific outcome measures, such as the VISA-G, which is not validated in Spanish. The WOMAC scale has been used to measure disability in patients with Greater Trochanteric Pain Syndrome (GTPS) who speak Spanish.
Hip Abduction Strength | From enrollment to the end of treatment at 4 months
  This will be defined as the amount of force measured by a manual dynamometer during a maximum voluntary isometric contraction. Strength is measured in kilograms (kg) using an Activforce 2 Dynamometer ACTVDIN® model. Participants will lie supine, with the test leg in an anatomical position at 0º hip rotation, and the opposite leg slightly flexed. The dynamometer will be positioned 5 cm proximal to the lateral malleolus, held externally by the examiner, who will stand on the same side as the tested leg. The contraction will be maintained for five seconds, and three measurements will be taken to obtain an average value. If compensatory movements are detected during a measurement, it will not be recorded, and another measurement will be taken.
Pain | From enrollment to the end of treatment at 4 months
  Participants will indicate their pain intensity on a 100 mm horizontal line, with "no pain"; at the far left (score 0) and "worst imaginable pain"; at the far right (score 10), in relation to the most intense pain episode experienced during daily activities. The Visual Analogue Scale (VAS) has been shown to effectively detect changes in pain, with a minimum clinically significant difference established at 13 mm.
Passive Hip Range of Motion | From enrollment to the end of treatment at 4 months
  It will be measured using an 18 cm plastic universal goniometer (Sammons Preston-Rolyan®). The following movements will be measured: flexion, extension, internal rotation, external rotation, and abduction until the end range without pain. Each movement will be measured three times, and the average value will be used in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

REFERENCES:
- [Background] Brennan KL, Allen BC, Maldonado YM. Dry Needling Versus Cortisone Injection in the Treatment of Greater Trochanteric Pain Syndrome: A Noninferiority Randomized Clinical Trial. J Orthop Sports Phys Ther. 2017 Apr;47(4):232-239. doi: 10.2519/jospt.2017.6994. Epub 2017 Mar 3. PMID 28257614
- [Background] Ceballos-Laita L, Jimenez-Del-Barrio S, Marin-Zurdo J, Moreno-Calvo A, Marin-Bone J, Albarova-Corral MI, Estebanez-de-Miguel E. Effectiveness of Dry Needling Therapy on Pain, Hip Muscle Strength, and Physical Function in Patients With Hip Osteoarthritis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):959-966. doi: 10.1016/j.apmr.2021.01.077. Epub 2021 Feb 7. PMID 33567336
- [Background] Fernandez-de-Las-Penas C, Nijs J. Trigger point dry needling for the treatment of myofascial pain syndrome: current perspectives within a pain neuroscience paradigm. J Pain Res. 2019 Jun 18;12:1899-1911. doi: 10.2147/JPR.S154728. eCollection 2019. PMID 31354339
- [Background] French HP, Woodley SJ, Fearon A, O'Connor L, Grimaldi A. Physiotherapy management of greater trochanteric pain syndrome (GTPS): an international survey of current physiotherapy practice. Physiotherapy. 2020 Dec;109:111-120. doi: 10.1016/j.physio.2019.05.002. Epub 2019 Jun 2. PMID 31493863
- [Background] Dieterich AV, Pickard CM, Strauss GR, Deshon LE, Gibson W, McKay J. Muscle thickness measurements to estimate gluteus medius and minimus activity levels. Man Ther. 2014 Oct;19(5):453-60. doi: 10.1016/j.math.2014.04.014. Epub 2014 May 10. PMID 24880207
- [Background] Schneider E, Moore ES, Stanborough R, Slaven E. Effects of Trigger Point Dry Needling on Strength Measurements and Activation Levels of the Gluteus Medius: A Quasi-Experimental Randomized Control Study. Int J Sports Phys Ther. 2022 Dec 1;17(7):1404-1416. doi: 10.26603/001c.55536. eCollection 2022. PMID 36518833
- [Background] Fearon AM, Scarvell JM, Neeman T, Cook JL, Cormick W, Smith PN. Greater trochanteric pain syndrome: defining the clinical syndrome. Br J Sports Med. 2013 Jul;47(10):649-53. doi: 10.1136/bjsports-2012-091565. Epub 2012 Sep 14. PMID 22983121
- [Background] Grimaldi A, Mellor R, Hodges P, Bennell K, Wajswelner H, Vicenzino B. Gluteal Tendinopathy: A Review of Mechanisms, Assessment and Management. Sports Med. 2015 Aug;45(8):1107-19. doi: 10.1007/s40279-015-0336-5. PMID 25969366
- [Background] Hilligsoe M, Rathleff MS, Olesen JL. Ultrasound Definitions and Findings in Greater Trochanteric Pain Syndrome: A Systematic Review. Ultrasound Med Biol. 2020 Jul;46(7):1584-1598. doi: 10.1016/j.ultrasmedbio.2020.03.008. Epub 2020 May 5. PMID 32381380
- [Background] Plinsinga ML, Ross MH, Coombes BK, Vicenzino B. Physical findings differ between individuals with greater trochanteric pain syndrome and healthy controls: A systematic review with meta-analysis. Musculoskelet Sci Pract. 2019 Oct;43:83-90. doi: 10.1016/j.msksp.2019.07.009. Epub 2019 Jul 25. PMID 31369906
- [Background] Segal NA, Felson DT, Torner JC, Zhu Y, Curtis JR, Niu J, Nevitt MC; Multicenter Osteoarthritis Study Group. Greater trochanteric pain syndrome: epidemiology and associated factors. Arch Phys Med Rehabil. 2007 Aug;88(8):988-92. doi: 10.1016/j.apmr.2007.04.014. PMID 17678660
- [Background] Lespasio MJ. Lateral Hip Pain: Relation to Greater Trochanteric Pain Syndrome. Perm J. 2022 Jun 29;26(2):83-88. doi: 10.7812/TPP/21.110. Epub 2022 Jun 15. PMID 35933677
- [Background] (1) Fredericson M, Lin CY, Chew K. Greater Trochanteric Pain Syndrome. Essentials of Physical Medicine and Rehabilitation 2021 -02-27:346.
- [Background] Grimaldi A, Mellor R, Nicolson P, Hodges P, Bennell K, Vicenzino B. Utility of clinical tests to diagnose MRI-confirmed gluteal tendinopathy in patients presenting with lateral hip pain. Br J Sports Med. 2017 Mar;51(6):519-524. doi: 10.1136/bjsports-2016-096175. Epub 2016 Sep 15. PMID 27633027